CLINICAL TRIAL: NCT01484886
Title: Prospective Randomized Controlled Clinical Trial Comparing a Restrictive Versus Liberal Transfusion Strategy in Neonates and Infants Undergoing Surgery for Congenital Heart Disease
Brief Title: Restrictive Versus Liberal Transfusion Protocol in Infants Undergoing Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, jill cholette, Assistant Professor of Pediatrics, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 38569
Record Dates: First submitted 2011-11-12; First posted 2011-12-02 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-09

CONDITIONS: Impaired Oxygen Delivery; Congenital Heart Disease
Keywords: Hemoglobin; Congenital heart disease; Cardiac surgery; Red blood cell transfusion; Number of red blood cell transfusions
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Erythrocyte Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Restrictive transfusion strategy (Experimental): RBC will be transfused if the hemoglobin level falls below 7 for bi-ventricular repairs and under 9.0 for single ventricle palliations.
  Interventions: Other: Red blood cell transfusion
- Liberal RBC transfusion strategy (Experimental): RBCs will be transfused for Hemoglobin under 9.5 for biventricular repairs and under 12 for single ventricle palliations.
  Interventions: Other: Red blood cell transfusion

INTERVENTIONS:
Other: Red blood cell transfusion — 10cc/kg weight RBC transfusion as needed according to hemoglobin level
Other: Red blood cell transfusion — 10cc/kg body weight RBC will be transfused for hemoglobin under 9.5 for biventricular repairs and under 12 for single ventricle palliations.
  Arms: Liberal RBC transfusion strategy

SUMMARY:
In neonates and infants </= 10 kg following cardiac surgery for congenital heart disease a more restrictive red blood cell (RBC) transfusion strategy will be as effective as, and possibly superior to, a liberal RBC strategy. Allowing lower hemoglobin concentration will not affect the cardiac or pulmonary status of the patient.

ELIGIBILITY:
Inclusion Criteria:

* children </= 6 months of age with congenital cardiac disease undergoing cardiac surgery with cardiopulmonary bypass.

Exclusion Criteria:

* presence of a known bleeding disorder or coagulopathy.
* age > 6 months,
* lack of informed consent.

Max Age: 7 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 162 (Actual)
Dates: Start 2012-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
oxygen utilization derived from the arterio-venous oxygen difference. | 3 days
  Arterial and venous oxygen saturations will be measured every four hours x 48-72 hours and will be used to calculate arterio-venous oxygen content differences.

SECONDARY OUTCOMES:
volume of RBC transfused | 7 days
  The total numbers of RBC transfusions given during the immediate post-op period (1st 7 days) will be compared between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States